CLINICAL TRIAL: NCT02852148
Title: A Prospective, Non-comparative, Multicentre Study to Evaluate a Silver Coated Antimicrobial Barrier Wound Dressing (ACTICOAT™) in the Treatment of Burns and Chronic Wounds.
Brief Title: ACTICOAT™ for the Treatment of Burns and Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1601ACT
Record Dates: First submitted 2016-06-24; First posted 2016-08-02 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Wounds and Injuries; Burns; Pressure Ulcer; Foot Ulcer
Keywords: Wound; Pressure Ulcer; Diabetic Foot Ulcer; Venous Leg Ulcer; Burn; Quality of Life
MeSH Terms: conditions — Wounds and Injuries; Burns; Pressure Ulcer; Foot Ulcer; Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACTICOAT (Experimental): ACTICOAT is a silver coated antimicrobial barrier dressing. ACTICOAT dressings consist of three layers: an absorbent inner core of polyester and rayon sandwiched between outer layers of silver coated, low adherent, high density polyethylene mesh.
  Interventions: Device: ACTICOAT

INTERVENTIONS:
Device: ACTICOAT — ACTICOAT is a silver coated antimicrobial barrier dressing. ACTICOAT dressings consist of three layers: an absorbent inner core of polyester and rayon sandwiched between outer layers of silver coated, low adherent, high density polyethylene mesh.

SUMMARY:
The aim of the study is to evaluate participant reported quality of life, safety, and overall performance with ACTICOAT in a clinical setting.

DETAILED DESCRIPTION:
ACTICOAT is a silver coated antimicrobial barrier wound dressing for the treatment of a variety of wound types. It is widely used in routine clinical practice within the UK. ACTICOAT is CE marked and will be used within the intended indications for use. The proposed study is required for regulatory purposes.

Primary Objective: To evaluate change in health related quality of life, associated with treatment. The primary outcome measure / endpoint will be change in EQ-5D 5L mean single index utility scores from baseline to 3 weeks.

The study will also seek to gather and report relevant safety and performance data and evaluate change, where applicable, for outcomes including: clinical signs and symptoms of infection; wound length / width / depth; wound healing measures; tissue staining; pain, adherence, and pain on application / removal; wear time; adverse events and device deficiencies.

In total 25 participants will be recruited into the trial, comprising a minimum of 8 participants with a full or partial thickness burn and a minimum of 8 participants with a full or partial thickness chronic wound. All participants will have their wound dressed using ACTICOAT, and will be followed-up for 3 weeks.

ELIGIBILITY:
INCLUSION CRITERIA

1. Must provide informed consent to participate in the study.
2. Eighteen (18) years of age or older.
3. Males and females.
4. Able to follow instructions and be deemed capable of completing the EQ-5D 5L Questionnaire appropriately.
5. Willing and able to make all required study visits, and provide a daytime telephone number on which they can be contacted directly.
6. Presenting with either a chronic wound or burn which is deemed suitable for treatment with ACTICOAT and meets either of the following requirements:

   1. A full or partial thickness chronic (≥ 4 weeks duration) wound, consisting of a Venous Leg Ulcer, Pressure Ulcer or Diabetic Foot Ulcer, which in the opinion of the Investigator, or delegated Sub-Investigator, appears to be infected based on documented clinical signs and symptoms of infection.
   2. A recently acquired (≤ 7 days) non-infected burn, comprising a full or partial thickness wound, covering a minimum 0.5% TBSA. The maximum must be less than 10% TBSA. Absence of infection will be determined by the Investigator / Sub-Investigator.

EXCLUSION CRITERIA

1. Contraindications or hypersensitivity to the use of the test article, ancillary products or their components (e.g., known sensitivity to silver).
2. Participation in the treatment period of another clinical trial within thirty (30) days of Visit 1.
3. Treatment with any other silver dressing (i.e. non ACTICOAT dressing) within seven (7) days of Visit 1.
4. Patients with skin features which in the opinion of the Investigator, will interfere with the study assessments.
5. Patients requiring concomitant use of NPWT on the reference wound.
6. Patients who have participated previously in this clinical trial and who have healed or been withdrawn.
7. Patients with a history of poor compliance with medical treatment.
8. Patients who, in the opinion of the Investigator, are experiencing burn shock.
9. Patients with any other medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Change in EQ-5D 5L mean single index utility scores (EuroQol Research Foundation 2015). | 21 days

SECONDARY OUTCOMES:
Clinical signs and symptoms of infection | 21 days
  Wound infection checklist. Simple checklist consisting of thirteen separate 'observable signs of critical colonisation or infection at the reference wound', namely: 'Wound static or deteriorating'; 'Increased exudate/secretion levels'; 'Increased temperature around wound'; 'Discoloration of granulation tissue'; 'Increased pain'; 'Tissue necrosis'; 'Oedema'; 'Dehiscence'; 'Friable granulation'; 'Local erythema'; 'Purulent drainage'; 'Odour'; 'Other'. Total scale score = the sum of checked items, ranging from 0 to 13
Wound length | 21 days
Wound width | 21 days
Wound depth | 21 days
Reference wound healed (% re-epithelialized) | 21 days
Amount of healthy tissue (% tissue types) | 21 days
Condition of surrounding skin | 21 days
  Condition of surround skin checklist. Simple checklist consisting of six items used to document the 'condition of the surrounding skin' around the wound, namely: 'Healthy'; 'Fragile'; 'Inflamed'; 'Macerated'; 'Dry and flaky'; 'Other'. No summation of items
Extent of tissue staining | 21 days
  Tissue staining checklist. Simple checklist for documenting any observed instances and 'Extent of tissue staining' following use of the dressing, and consisting of four items, namely: 'None'; 'Slight'; 'Moderate'; and 'Extensive'. No summation of items
Pain on dressing application | 21 days
  Pain/stinging Likert scale for dressing application. Eleven point Likert scale for use in recording 'Level of pain/stinging experienced by the subject on application of the ACTICOAT dressing(s)', ranging from 0 (no pain/stinging) to 10 (extreme pain/stinging)
Pain on dressing removal | 21 days
  Pain Likert scale for dressing removal. Eleven point Likert scale for use in recording 'Level of pain experienced by the subject on removal of the ACTICOAT dressing(s)', ranging from 0 (no pain) to 10 (extreme pain).
Ease of dressing application | 21 days
  Ease of dressing application question. Single item asking 'Was it easy to apply the ACTICOAT dressing(s)?', with a simple response format of 'Yes' or 'No - please give reason', accompanied by a further free text response option for reason(s) why the dressing was not easy to apply
Ease of dressing removal | 21 days
  Ease of dressing removal question. Single item asking 'Was the ACTICOAT dressing easy to remove?', with a simple response format of 'Yes' or 'No - please explain', accompanied by a further free text response option for reason(s) why the dressing was not easy to remove
Serious adverse events | 21 days
  Record of absolute number of serious adverse events observed in the study, together with associated details
Non-serious adverse events | 21 days
  Record of the absolute number of non-serious adverse events observed in the study, together with associated details
Device deficiencies | 21 days
  Record of the absolute number of device deficiencies observed in the study, together with associated details

CONTACTS AND LOCATIONS:
Overall Officials: Beate Hanson, VP, PhD, Study Chair — Smith & Nephew, Inc.; Lyn Wilson, MA, Principal Investigator — Pinderfield Hospitals
Locations (3):
- United Kingdom (3):
  - Northumbria Healthcare NHS Foundation Trust, Ashington
  - Leeds Wounds Research Unit, Leeds
  - The Mid Yorkshire Hospitals NHS Trust, Wakefield

IPD SHARING:
Plan to Share IPD: No